CLINICAL TRIAL: NCT06332248
Title: A Double-blind, Randomized Placebo-controlled Intervention Study About Possible Effects of the Dietary Supplement Magnesium.
Brief Title: Possible Effects of the Dietary Supplement Magnesium Compared to Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dan Hasson (Other)
Collaborators: Stiftelsen Stressmottagningen (Unknown); AFA Insurance (Industry)
Responsible Party: Sponsor-Investigator, Dan Hasson, PhD, Associate Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014/1023-31/4 & 2014/274-31/5
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Health Promotion
Keywords: Self-rated health; Stress; Magnesium supplement; Placebo; Double-blind; Randomized controlled trial (RCT); Wellbeing; Recovery; Stress management
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Intervention Model Description: Participants received either 375 mg nutritional supplement magnesium or placebo pill.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium 375 mg (Experimental): 375 mg dietary supplement magnesium, one pill daily for up to 3 months.
  Interventions: Dietary Supplement: Magnesium
- Placebo (Placebo Comparator): Placebo (rice powder), one pill daily for up to 3 months. Identical appearance as the magnesium pill.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium — The dietary supplement magnesium (375 mg) was given daily for up to 3 months (oral intake).
  Arms: Magnesium 375 mg
Dietary Supplement: Placebo — Placebo tablet, oral intake once a day for up to three months.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial was to investigate possible outcomes of the nutritional supplement magnesium compared to placebo in healthy, working adults. The main questions it aimed to answer were:

* Are there differences in ratings of health, stress, well-being and work environment indicators between individuals intaking 375 mg magnesium (daily for 3 months) compared to placebo?
* Are there differences in hearing, measured with hearing tests between those receiving 375 mg magnesium compared to placebo?

Participants were asked to ingest 375 mg magnesium or placebo daily for 3 months.

Researchers compared the group ingesting magnesium with the group ingesting placebo pills to see if there were any differences in for example self-rated health, recovery, wellbeing, etc.

DETAILED DESCRIPTION:
Summary: The aim of the sub-study was to investigate possible beneficial effects of magnesium as a nutritional supplement regarding self-reported health, ill-health, pain, hearing, fatigue, signs of long term stress and more. The study was designed as a double-blind placebo-randomized controlled study, meaning that each enrolled individual was randomized to either 375 mg magnesium or placebo pills. Clinical hearing tests, blood pressure, pulse and creatinine were conducted and collected. Extensive questionnaires were distributed at baseline (T1) and after approximately 3 months (T2) of daily pill intake in order to evaluate possible effects. All participants were adults and healthy enough to work.

Previous research studies have shown that magnesium has promising effects to counteract or mitigate for instance headache/migraine, muscle cramps, high blood pressure, asthma as well as hearing problems such as tinnitus and sound sensitivity (hyperacusis). Magnesium deficiency is related to reduced immune function and physical symptoms such as migraine, muscle cramps, osteoporosis and high blood pressure/metabolic syndrome.

Magnesium is one of the body's most common and important minerals. It is involved in the regulation of the nerve activity and the muscle function. As a dietary supplement, it is affordable, easily administrated and safe. Adverse effects in the form of diarrhea can occur if magnesium is greatly overdosed. The participants in this trial were informed about this and possible other adverse effects and were recommended to terminate participation or decrease the intake (e.g., take half a pill) in case of any experienced adverse effects. They were also encouraged to report any adverse effects immediately.

The primary objective with the study was to investigate if there were differences between the treatment group (magnesium) and the control group (placebo) over time in health-related outcomes, recovery and well-being.

The present study was conducted as a separate study within a larger intervention study for employees at 21 schools in Stockholm, Sweden. The purpose of the larger intervention study was to evaluate possible effects of systematic interventions for health promotion and work environment improvements, as well as to counteract harmful stress and long-term sick-leave.

Employees could choose to participate in the larger intervention study, the sub study about magnesium/placebo, both or none of them.

Individuals enrolled in the magnesium/placebo randomized control trial by signing up for a session of hearing tests and other physiological measures approximately one week before the session. The researchers randomized each enrolled individual and prepared a kit containing the randomized jar of pills (magnesium or placebo), a paper adherence calendar, general information about the study along with instructions for intake and a protocol used by the researchers during the session. In some cases, there were some last-minute enrollments who were randomized onsite. During the session (at the participants workplace), hearing tests were performed with portable equipment, and measures of blood pressure, pulse and creatinine were performed. At the end of the session, the participant was provided with the magnesium/placebo kit and was asked to fill out a web-based questionnaire. The same measures were performed after approximately three months, except for the creatinine test. Participants were also asked to fill out another web-based questionnaire and were asked to return the magnesium/placebo kit and the compliance calendar.

ELIGIBILITY:
Inclusion Criteria:

Individuals employed at the participating organizations (21 schools and one white collar organization) who provided their informed consent and were at least 18 years old.

Exclusion Criteria:

1. Individuals with creatinine levels more than195 μmol/L for women and more than 230 μmol/L for men.
2. Individuals who had undergone a liver transplant.
3. Lithium intake or prescription.

Pregnant women were disadvised from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2015-05-28 (Actual)

PRIMARY OUTCOMES:
Time x group difference in HealthWatch-11 (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  The questionnaire HealthWatch-11 (HW-11) was utilized with all 11 items: self-rated health, sleep, concentration ability, stress, energy level, control, social support, work efficiency, job satisfaction, workload and work atmosphere. Scale type is verbal rating scale (VRS) for all items (stress and work efficiency use visual analogue scale). The minimum value is 0 and the maximum value is 100 for all items. Higher values mean better outcomes for all variables except for stress and workload, where lower values are better and higher values are worse.

SECONDARY OUTCOMES:
Intervention compliance measure 1 (objective, number of pills left) | From Baseline to the end of intervention at approximately 3 months.
  Compliance in the intervention was assessed by counting the number of pills left in the jar. Each jar contained 100 pills at baseline.
Intervention compliance measure 2 (subjective, marked days in calendar) | From Baseline to the end of intervention at approximately 3 months.
  Compliance in the intervention was assessed by counting the number of marked days in the compliance calendar.

OTHER OUTCOMES:
Time x group difference in Oldenburg Burnout Inventory (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  The questionnaire Oldenburg Burnout Inventory (OLBI) was utilized with 10 items to assess signs of emotional exhaustion and disengagement. Scale type is Likert with 4 steps where the minimum value is 1 and the highest 4. Higher values are worse than lower values (4 items are reversed in coding).
Time x group difference in Karolinska Sleep Questionnaire | From Baseline to the end of intervention at approximately 3 months.
  The questionnaire Karolinska Sleep Questionnaire (KSQ) was utilized with 13 items to assess 3 aspects of sleeping problems. Scale type is Likert with 5 steps (minimum value 0 and maximum value 5) where lower values are better and higher values are worse.
Time x group difference in Pure Tone Audiogram (clinical hearing test) | From Baseline to the end of intervention at approximately 3 months.
  The hearing test Pure tone audiogram (PTA) was conducted to establish thresholds for hearing in the frequencies 125 hertz (Hz), 250 Hz, 500 Hz, 1000 Hz, 2000 Hz, 3000 Hz, 4000 Hz, 6000 Hz and 8000 Hz. The tests were conducted on each ear separately.
Time x group difference in Speech in noise test (clinical hearing test) | From Baseline to the end of intervention at approximately 3 months.
  This test was conducted in order to assess hearing in noisy environments. The participant was first asked to establish the Most Comfortable Loudness level (MCL), this was done on one ear only. MCL was established by the participant listening to a recorded male voice saying monosyllabic words in Swedish. The examiner adjusted the loudness level based on the participants' instructions in 5 decibel (dB) steps. Once MCL was established, the speech in noise test was started. The examiner played at set of 25 words per ear with a background noise that was 10 dB lower than the volume of the words. The participant was asked to repeat the words as they heard them. The examiner marked the answers as correct or incorrectly repeated. More correctly repeated words were considered better and more incorrectly repeated words worse. The participant's age is also taken into account since the ability to hear words in a noisy environment declines with age.
Time x group difference in Uncomfortable loudness level (clinical hearing test) | From Baseline to the end of intervention at approximately 3 months.
  Uncomfortable loudness level (UCL) is a test to assess possible sensitivity to sound (hyperacusis). The participant was instructed that they would be hearing a man's voice saying words and that the examiner would increase the volume until the participant experienced the loudness level to start being uncomfortably loud. The maximum sound level was 110 decibel (dB).
Time x group difference in single questionnaire item assessing sick leave | From Baseline to the end of intervention at approximately 3 months.
  The single item "About how many days have you been on sick leave or reported in sick during the past 12 months?" was utilized to assess sick leave. Responses were given on a 5 point Likert scale ranging from 1 to 5, where 1 was better (no sick leave) and 5 was worse (91 days or more of sick leave).
Time x group difference in single questionnaire item assessing sickness presenteeism | From Baseline to the end of intervention at approximately 3 months.
  The single item "How many times during the past 12 months have you gone to work despite that you thought you should have been on sick-leave considering your health status?" was utilized to assess sickness presenteeism. Responses were given on a 4 point Likert scale ranging from 1 to 4 where 1 was better (None) and 4 was worse (4 times or more).
Time x group difference in prevalence of pain (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  Prevalence of pain was assessed using a Likert scale (1=Yes and 0=No). The following 8 body areas were assessed: head, neck, shoulder, arm/hand, upper back, lower back, legs and general pain.
Time x group difference in pain frequency (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  The frequency of pain was assessed utilizing a 4 point Likert scale ranging from 1 to 4 where lower values were better than higher values.
Time x group difference in pain discomfort (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  Pain discomfort was assessed utilizing a Visual Analogue Scale (VAS) ranging from 1 to 100 where lower values were better (less discomfort) than higher values (more discomfort).
Time x group difference in pain intensity (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  Pain intensity was assessed utilizing a Visual Analogue Scale (VAS) ranging from 1 to 100 where lower values were better (lower intensity) than higher values (higher intensity).
Time x group difference in functional impairment due to pain (questionnaire) | From Baseline to the end of intervention at approximately 3 months.
  Functional impairment due to pain was assessed using a Likert scale (1 = Yes and 0 = No) where higher values are worse. Functional impairment was assessed in the following 3 areas: difficulties to carry out your everyday chores due to pain, difficulties to sleep due to pain and difficulties to carry out your work due to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hasson, PhD, Principal Investigator — Karolinska Institutet and Mayo Clinic

IPD SHARING:
Plan to Share IPD: No